CLINICAL TRIAL: NCT06277089
Title: Curve Correction of Early Onset Scoliosis by Mehta Serial Casts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Kamal Zohery, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Correction of EOS by casts
Record Dates: First submitted 2024-01-13; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Casts, Surgical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Correction of EOS by serial cast (Other)
  Interventions: Other: Casts

INTERVENTIONS:
Other: Casts — According to level of scoliosis cast done and recast in a serial manner

SUMMARY:
Assessment of the role of Mehta Serial Casts in Curve Correction of Early Onset Scoliosis

DETAILED DESCRIPTION:
Early Onset Scoliosis refers to various types of Scoliosis with onset before 10 years of age .In addition to spinal Deformity Progressive Scoliosis will also affect the development of thoracic cage and lungs . So Early correction is important .

Curve correction can done by operative and nonoperative techniques . Our Study include the curve correction by Mehta Serial Casts which not need for blood transfusion and has a good role in stop progression and delay the need for surgery .

ELIGIBILITY:
Inclusion Criteria:

* All cases with Early Onset Scoliosis up to 10 years Age presenting to Assiut University Hospitals during 2 years period .

Exclusion Criteria:

* Cases with previous spine surgery and those whose guardians refuse to participate in the study .

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference of the scoliotic cobb angle at last cast | 1 year
  Measurement of Cobb angle in every visit and find the difference of the Scoliotic Cobb angle between first and last visit to assist the Correction ( Cobb angle measured by X Ray

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Mostafa El Sharkawi, Study Director — Prof.dr; Nariman Elsayed Mohammad ABOL Oyoun, Study Director — Prof.dr

REFERENCES:
- [Background] Thorsness RJ, Faust JR, Behrend CJ, Sanders JO. Nonsurgical Management of Early-onset Scoliosis. J Am Acad Orthop Surg. 2015 Sep;23(9):519-28. doi: 10.5435/JAAOS-D-14-00019. PMID 26306805
- [Background] Matsumoto H, Auran E, Fields MW, Hung CW, Hilaire TS, Roye B, Sturm P, Garg S, Sanders J, Oetgen M, Levine S, Roye D, Vitale M; Pediatric Spine Study Group. Serial casting for early onset scoliosis and its effects on health-related quality of life during and after discontinuation of treatment. Spine Deform. 2020 Dec;8(6):1361-1367. doi: 10.1007/s43390-020-00175-5. Epub 2020 Aug 5. PMID 32757176
- [Background] Mahajan R, Kishan S, Mallepally AR, Shafer C, Marathe N, Chhabra HS. Evolution of casting techniques in early-onset and congenital scoliosis. J Clin Orthop Trauma. 2020 Sep-Oct;11(5):810-815. doi: 10.1016/j.jcot.2020.06.034. Epub 2020 Jul 8. PMID 32879567